CLINICAL TRIAL: NCT03382769
Title: Hearing Loss in Older Adults: A Randomized Controlled Trial of Immediate Versus Delayed Cochlear Implantation.
Brief Title: Hearing Loss in Older Adults Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early terminated due to COVID-19 public health emergency, with a patient population in vulnerable populations (older adults) seeking cochlear implantation as elective Standard of Care.
Sponsor: Cochlear (Industry)
Collaborators: CogState Ltd. (Industry); Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5693
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss, Bilateral
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Bilateral | interventions — Cochlear Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A (Immediate Cochlear Implantation) (Experimental): Group A will consist of 30 individuals who are candidates for cochlear implantation. They will be unilaterally implanted immediately after initial study testing has been completed and then be followed for 12 months after device activation.
  Interventions: Device: Cochlear implantation
- Group B (Delayed Cochlear Implantation) (Active Comparator): Group B will consist of 30 individuals who are candidates for cochlear implantation. They will continue to wear hearing aids after enrolling in the study and then be unilaterally implanted 6 months after enrollment and followed for 6 more months after device activation.
  Interventions: Device: Cochlear implantation

INTERVENTIONS:
Device: Cochlear implantation — Unilateral implantation with a commercially approved Nucleus cochlear implant

SUMMARY:
This is a prospective, 1:1 randomized controlled trial of immediate versus delayed cochlear implantation (CI) on hearing handicap, communicative function, loneliness, mental wellbeing, and cognitive functioning. Participants are randomized 1:1 to an immediate cochlear implant intervention group versus a hearing aid control intervention.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling
* Proficient in English
* Oral communicator
* PTA (500, 1000 & 2000 Hz) ≥ 70 dB HL hearing loss duration ≥1 and no more than 30 years
* Active daily hearing aid users
* HHIE-S score greater than or equal to 24
* MoCA score greater than or equal to 20
* Post-linguistic onset sensorineural hearing loss and meet applicable FDA and/or Medicare candidacy criteria for cochlear implantation
* Willing to consent for the study, to be randomized to either group, to utilize bimodal hearing for the duration of the trial (if clinically appropriate), and follow the study protocol

Exclusion Criteria:

* Prelingual or perilingual severe-to-profound hearing loss
* Previous cochlear implantation in either ear
* Hearing loss of neural or central origin
* Permanent conductive hearing impairment (e.g. otosclerosis)
* Medical, audiological, or psychological conductions that might contraindicate participation in the clinical investigation
* Self reported disability in 2 or more activities of daily living
* Vision impairment worse than 20/40 on a near vision card

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2020-01-04 (Actual); Study Completion 2020-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David N Cade, MD, MBA, Study Director — Cochlear
Locations (8):
- United States (8):
  - Arizona Center for Neurosciences, Tucson, Arizona
  - House Ear Institute, Los Angeles, California
  - Washington University, St Louis, Missouri
  - New York Eye and Ear Infirmary of Mount Sinai, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - University of Cincinnati Health, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A (Immediate Cochlear Implantation) | Group B (Delayed Cochlear Implantation)
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Study terminated due to COVID 19
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Immediate Cochlear Implantation) | Group B (Delayed Cochlear Implantation) | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Hearing Handicap
Description: The SSQ-12 is comprised of 12 items using the response format on a scale from 0 to 10, were 0 equals no ability and 10 equals perfect ability. These are divided into three sub-scales and the questions 1-5 are from the speech sub-scale, 6-8 from the spatial, and 9-12 from the qualities sub-scale. The three sub-scales are the average of the questions within. A 'not applicable' option is given for each item.
  Assessment of the impact of cochlear implantation versus continued hearing aid is then calculated and the theoretical score could vary between -10 to + 10. The higher the score the better benefit and positive score indicates improved hearing, a negative value an impaired hearing.
Time Frame: 6 months after enrollment
Population: Data was not collected as the study was terminated due to COVID-19
Arm/Group | Group A (Immediate Cochlear Implantation) | Group B (Delayed Cochlear Implantation)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: All Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed although there was 1 subject enrolled and withdrawn due to not meeting candidacy requirements and study was terminated due to COVID 19.
Arm/Group | Group A (Immediate Cochlear Implantation) | Group B (Delayed Cochlear Implantation)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT03382769/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT03382769/SAP_001.pdf